CLINICAL TRIAL: NCT05272735
Title: HBV Vaccination of Healthy Volunteers to Evaluate the Composition of Germinal Centers
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Rockefeller University (Other)
Collaborators: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GVI 1028
Record Dates: First submitted 2022-02-28; First posted 2022-03-09 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Hepatitis B
MeSH Terms: conditions — Hepatitis B | interventions — Hepatitis B Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Hepatitis B Vaccine (Recombinant) (Experimental): Hepatitis B Vaccine (Recombinant) 20 mcg intramuscular injection at 0-1-6 months
  Interventions: Biological: Hepatitis B Vaccine (Recombinant)

INTERVENTIONS:
Biological: Hepatitis B Vaccine (Recombinant) — Hepatitis B Vaccine (Recombinant) 20 mcg intramuscular injection at 0-1-6 months

SUMMARY:
Antibodies are the primary mediators of the protection against infection provided by vaccination. Antibodies become most powerful after the B cells that produce them undergo an evolutionary process called affinity maturation, in which antibodies increase their ability to bind to their targets, and thus neutralize pathogens. Affinity maturation occurs in structures within secondary lymphoid organs (for example lymph nodes or tonsils) known as germinal centers. Germinal centers are well known to be triggered by the first dose of vaccines, generating affinity matured plasma cells (B cells that secrete antibody into serum) and memory B cells, which can be converted into plasma cells by booster doses of vaccine. However, it is not fully understood the extent to which memory B cells can return to germinal centers again upon vaccine boosting. Such return would be very important to allow B cells, for example, to adapt to emerging variants of viruses such as influenza or SARS-CoV-2. This study will involve acquiring samples of B cells from germinal centers that form in response to vaccination with the highly effective hepatitis B vaccine. These cells will be analyzed to determine what fraction of them are memory B cells that returned to germinal centers upon boosting, information that is key to knowledge of how vaccine boosters work. Understanding the "rules" that govern how and when memory B cells choose to return to germinal centers in an effective vaccine such hepatitis B could help efforts to develop effective vaccination against more challenging, rapidly mutating viruses, such as influenza, HIV, and hepatitis C.

DETAILED DESCRIPTION:
A feature of the immune system of critical importance is its ability to mount a much stronger antibody response the second time a pathogen or antigen is encountered (1). This property underlies the need for "booster" doses to ensure the effectiveness of vaccination. The booster effect derives in part from the generation, by the primary response, of expanded clones of memory B cells (MBCs). Upon re-exposure to antigen, MBCs rapidly proliferate and differentiate into plasma cells, generating high titers of serum antibody over a short period of time. Because most MBCs that respond to boosting have also undergone affinity maturation in germinal centers (GCs) during the primary response (2), MBC-derived antibody has both higher affinity and higher cross-variant breadth than primary antibody (3).

A common assumption in the vaccinology field has been that, in addition to forming plasma cells, MBCs will also generate secondary GCs upon boosting with high efficiency, allowing them to re-evolve their immunoglobulins to adapt to variant strains of a pathogen (4-6). This assumption forms the basis of multiple attempts to guide B cell clones towards broad reactivity to influenza or HIV by iteratively recruiting them to germinal centers by sequential immunization.

Recent work using genetic tracing of memory B cell clones in mice questions this assumption (7). Using fate-mapping of primary-GC-derived B cells, results showed that mouse MBCs are remarkably inefficient at forming secondary GCs, which instead consist predominantly (>90%) of cells derived from naïve precursors engaged only by the boost but not by the prime (2). Partly in contrast to the mouse findings, a recent study using fine-needle aspirates (FNA) to sample vaccine-draining lymph node GCs in healthy humans immunized with a quadrivalent influenza vaccine showed that MBC participation in recall GCs can vary depending on the individual sampled, ranging from approximately 5%, a proportion similar to that found in mice, to up to ~65% in one individual (8). This wide range was not recapitulated in our mouse models. A key unknown in this study was the degree of prior exposure of each individual to influenza antigens, via either infection or vaccination. Long histories of exposure can generate influenza-specific MBC compartments in blood that represent >1% of all B cells (9). On the other hand, simpler exposure regimens, such as HPV, tetanus, and HBV vaccination, generate much lower frequencies of antigen-specific MBCs, in the high tens to low hundreds per million B cells, comparable to frequencies found after single immunization or infection in mice (10-14).

There is a hypothesize that the wide range of MBC re-entry into recall GCs observed after human influenza vaccination reflects differences in the history of exposure of individuals to influenza antigens, rather than more fundamental differences in MBC biology between humans and mice. There is expectation the findings of this study will be of critical value to the general understanding of vaccination, as well as to those seeking to generate influenza and HIV broadly neutralizing antibodies (bNAbs) by vaccination. These studies will also be critical to determine the extent to which mouse models reliably predict human responses at the clonal level and can therefore be used to test sequential immunization regimens.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Age 18-50 years Note: The HBV vaccine dose will be adjusted according to the Package Insert for participants who are 18 and 19 years of age.
* No prior history of HBV infection or vaccination.

Exclusion Criteria:

* HBV seropositivity (e.g. HBsAb, HBcAb or HBeAb)
* HIV infection
* Chronic HCV infection
* Pregnancy or lactation
* History of allergic reaction to any components of the HBV vaccine
* History of significant local or systemic reactogenicity to vaccines (eg, anaphylaxis, respiratory difficulties, angioedema, injection site necrosis or ulceration)
* Any clinically relevant abnormality on history or examination, including history of immunodeficiency or autoimmune disease; use of systemic corticosteroids (the use of topical or inhaled steroids is permitted), immunosuppressive, anticancer, antituberculosis or other medications considered significant by the Investigator within the previous 6 months; Note: The following exceptions are permitted and will not exclude study participation: use of corticosteroid nasal spray for rhinitis, topical corticosteroids for an acute uncomplicated dermatitis; or a short course (duration of 10 days or less, or a single injection) of corticosteroid for a non-chronic condition (based on Investigator clinical judgment) at least 2 weeks prior to enrollment in this study
* Any clinically significant acute or chronic medical condition that is considered progressive or in the opinion of the Investigator makes the volunteer unsuitable for participation in the study
* Bleeding disorder that was diagnosed by a physician (eg, factor deficiency, coagulopathy or platelet disorder that requires special precautions)
* Laboratory abnormalities:

Platelets <125,000 cells/mm3 PT/INR >1.3 PTT > 2 x ULN

* Receipt of live attenuated or mRNA vaccine within the previous 30 days or planned receipt within 30 days after IP administration; or receipt of other vaccine within the previous 14 days or planned receipt within 14 days after IP administration
* Participation in another clinical trial of an investigational product currently, within the previous 3 months or expected participation during this study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-12-10 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The Effects of HBV Vaccine on Memory B Cells | 6 months
  The percentage of B cells in GCs triggered by the third dose of HBV vaccine that can derive from memory B cells.

SECONDARY OUTCOMES:
B Cell Response to the HBV Vaccination | 6 months
  The percentage and characterization of the clonal and cellular dynamics of the B cell response to the three-dose sequence of HBV vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel D. Victora, PhD, Principal Investigator — The Rockefeller University
Locations (1):
- The Rockefeller University, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mesin L, Schiepers A, Ersching J, Barbulescu A, Cavazzoni CB, Angelini A, Okada T, Kurosaki T, Victora GD. Restricted Clonality and Limited Germinal Center Reentry Characterize Memory B Cell Reactivation by Boosting. Cell. 2020 Jan 9;180(1):92-106.e11. doi: 10.1016/j.cell.2019.11.032. Epub 2019 Dec 19. PMID 31866068